CLINICAL TRIAL: NCT03669471
Title: Muscular and Functional Hop Test Performance in Femoroacetabular Impingement Syndrome Patients 6-30 Months Post Hip Arthroscopy - a Cross-sectional Study
Brief Title: Muscular and Functional Performance in FAIS Patients
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Lasse Ishøi, Principal Investigator, Hvidovre University Hospital
Other Study IDs: FAIS2018
Record Dates: First submitted 2018-09-07; First posted 2018-09-13 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FAIS group: Subjects who have had a hip arthroscopy for femoroacetabular impingement during the preceding 6-30 months
  Interventions: Other: Testing of performance

INTERVENTIONS:
Other: Testing of performance — The cross-sectional evaluation will involve assessment of:
  1. Hip muscle function
  2. Single leg jump performance
  3. Self-reported hip and groin function
  4. Evaluation of return to sport
  5. Evaluation of satisfaction regarding usual-care post-operative rehabilitation
  The exercise-based treatment will involve criteria-based physiotherapy aiming at improving muscle function around the hip and trunk.
  Other Names: Exercise-based treatment

SUMMARY:
Following hip arthroscopy for femoroacetabular impingement syndrome (FAIS) decreased hip muscle strength for adduction, extension, flexion, and external rotation including impaired functional performance have been observed. However, no studies are lacking on more demanding muscular and functional parameters such as hip muscle rate of force development and reactive strength index. Information on such muscular properties following hip arthroscopy for FAIS may help guide future planning of post-operative rehabilitation strategies.

This is a cross-sectional study with an embedded prospective non-randomized study. The aim of the cross-sectional study is to investigate hip muscle function and functional performance in patients who have undergone hip arthroscopy for FAIS during the preceding 6-30 months.

The aim of the prospective non-randomized study is to investigate the effect of a 12-week structured and supervised physiotherapy-led intervention aiming at improving hip muscular function on self-reported hip and groin function including hip muscle function and functional performance.

Forty-five subjects from the Capital Region with an age of 18-40, who have undergone a hip arthroscopy for FAIS during the last 6-30 months, will be included in the cross-sectional study. Additionally, all included subjects will be offered to take part in the prospective non-randomized study consisting of 12 weeks of supervised and structured physiotherapy-led treatment.

The below measures will be obtained at baseline, and at 12-weeks follow-up if subjects are included in the prospective study. All testing, and supervised physiotherapy-led treatment, will be performed at Hvidovre Hospital:

1. Hip muscle function
2. Single leg jump performance
3. Self-reported hip and groin function
4. Evaluation of return to sport
5. Evaluation of satisfaction regarding usual-care post-operative rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Male/female at the age of 18-40 years at the time of surgery
* Undergone hip arthroscopy for FAIS during the previous 6-30 months (surgical procedure: cam resection and labral surgery)
* Pre-operative cam morphology specified as an alpha angle ≥55°

Exclusion Criteria:

* Pre-surgery joint space width <3 mm
* Any of the following surgical procedures at any time: extra articular surgery of the hip joint (except capsular closure), microfracture, periacetabular osteotomy, and surgery of the ligamentum teres; previous hip arthroscopy in the same hip joint; previous hip pathology such as Perthes' disease, slipped upper femoral epiphysis, hip dysplasia (Lateral Center Edge Angle <25°), and/or avascular necrosis; Any rheumatoid disease in the hip joint such as synovial chondromatosis.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects who have undergone hip arthroscopy for femoroacetabular impingement syndrome during the preceding 6-30 months in the Greater Copehangen Area
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Peak force | Baseline (week 0)
  Peak isometric hip torque (Nm/kg) of abduction, adduction, extension, and flexion
Rate of force development | Baseline (week 0)
  0-100 ms and 0-200 ms rate of torque development (Nm/s/kg) of abduction, adduction, extension, and flexion
Self-reported hip and groin function (subjects included in prospective study) | Baseline (week 0) and follow-up (week 12)
  Obtained using the Copenhagen Hip and Groin Outcome Score (HAGOS); Scale from 0 (extreme hip and groin problems) to 100 (no hip and groin problems)

SECONDARY OUTCOMES:
Single leg jump performance | Baseline (week 0)
  Reactive strength index obtained during a single leg drop jump test
Self-reported hip and groin function | Baseline (week 0)
  Obtained using the Copenhagen Hip and Groin Outcome Score (HAGOS); Scale from 0 (extreme hip and groin problems) to 100 (no hip and groin problems)
Return to sport | Baseline (week 0)
  Obtained using a return to sport questionnaire; Scale: Preinjury sport at preinjury level vs. not preinjury sport at preinjury level.
Satisfaction regarding usual-care post-operative rehabilitation | Baseline (week 0)
  Obtained using a questionnaire; Scale: Satisfied with regular post-operative rehabilitation vs. not satisfied with post-operative rehabilitation.
Change in Peak force (subjects included in prospective study) | Baseline (week 0) and follow-up (week 12)
  Peak isometric hip torque (Nm/kg) of abduction, adduction, extension, and flexion
Change in rate of force development (subjects included in prospective study) | Baseline (week 0) and follow-up (week 12)
  0-100 ms and 0-200 ms rate of torque development (Nm/s/kg) of abduction, adduction, extension, and flexion
Change in Single leg jump performance (subjects included in prospective study) | Baseline (week 0) and follow-up (week 12)
  Reactive strength index obtained during a single leg drop jump test

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Ishøi, Principal Investigator — Sports Orthopedic Research Center - Copenhagen (SORC-C), Ortopædkirurgisk Afdeling, Hvidovre Hospital
Locations (1):
- Testing and exercise-based intervention will be conducted at Hvidovre Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided